CLINICAL TRIAL: NCT01109199
Title: A Randomized, Double Blind, Placebo Controlled Trial Evaluating the Effects of a High Viscosity Dietary Fibre (PGX) Supplementation of a Low Calorie Diet on Appetite and Body Weight, in Overweight and Moderately Obese Females
Brief Title: Effects of a Dietary Fibre Supplementation of a Low Calorie Diet on Appetite and Body Weight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Center for Functional Medicine (Other)
Collaborators: University of British Columbia (Other); InovoBiologic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGX RCT Study
Record Dates: First submitted 2010-04-20; First posted 2010-04-23 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Appetite Suppression; Weight Loss
Keywords: viscous; fibre; polysaccharide; appetite; hunger; satiety; weight management
MeSH Terms: conditions — Weight Loss | interventions — PolyGlycoplex; Flour

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- PolyGlycopleX (PGX) (Experimental)
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- Rice Flour (Placebo Comparator)
  Interventions: Dietary Supplement: Rice flour

INTERVENTIONS:
Dietary Supplement: PolyGlycopleX (PGX) — The full dose of the study intervention is 15 grams per day and total number of calories with the LCD is 1000 kcal/day.
  Arms: PolyGlycopleX (PGX)
Dietary Supplement: Rice flour — The full dose of the placebo comparator is 15 grams per day and total number of calories with the LCD is 1000 kcal/day.
  Arms: Rice Flour

SUMMARY:
This 18 week, randomized, double blind, placebo controlled trial will examine the effects of thick dietary fibre (PGX) supplementation of a low calorie diet (LCD) on appetite, weight loss, body composition, and compliance in overweight and moderately obese female.

The investigators believe that 15 grams/day PGX supplementation of a low calorie diet over a 14-weeks period will elicit a better appetite score (e.g. reduced hunger) compared to the rice flour supplementation of the LCD.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 - 35 Kg/m2

Exclusion Criteria:

* Medications and supplements that affect appetite
* Known diabetes
* Contraindications to LCD
* Any other medical, social or geographic condition, which, in the opinion of the investigator would not allow safe completion of the protocol.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The difference in appetite score assessed from appetite Visual Analog Scale | 18 weeks

SECONDARY OUTCOMES:
Change in weight (kilograms) | 18 weeks
Change in percentage of body fat | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Lyon, M.D., Principal Investigator — Canadian Center for Functional Medicine
Locations (1):
- Canadian Center for Functional Medicine, Coquitlam, British Columbia, Canada